CLINICAL TRIAL: NCT05609370
Title: A Phase 1b/2, Randomized, Open-Label Study Investigating the Efficacy and Safety of LBL-007 Plus Tislelizumab in Combination With Bevacizumab Plus Fluoropyrimidine Versus Bevacizumab Plus Fluoropyrimidine as Maintenance Therapy in Patients With Unresectable or Metastatic Microsatellite Stable/Mismatch Repair Proficient Colorectal Cancer
Brief Title: A Study Investigating the Efficacy and Safety of LBL-007 Plus Tislelizumab in Combination With Bevacizumab Plus Fluoropyrimidine Versus Bevacizumab Plus Fluoropyrimidine in Participants With Unresectable or Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-LBL-007-201; CTR20223077 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2022-10-20; First posted 2022-11-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Unresectable or Metastatic Microsatellite Stable/Mismatch Repair Proficient Colorectal Cancer
Keywords: Colorectal Cancer; Microsatellite Stable; Mismatch Repair Proficient; Maintenance Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; Bevacizumab; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Phase 1b: Cohort -1: LBL-007 + Tislelizumab + Bevacizumab + Capecitabine (Experimental): LBL-007 (low dose) + tislelizumab (low dose once every 3 weeks) + bevacizumab (7.5 mg/kg once every 3 weeks) + capecitabine
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: Capecitabine
- Phase 1b: Cohort 1a: LBL-007 + Tislelizumab + Bevacizumab + Capecitabine (Experimental): LBL-007 (medium dose) + tislelizumab (low dose once every 3 weeks) + bevacizumab (7.5 mg/kg once every 3 weeks) + capecitabine
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: Capecitabine
- Phase 1b: Cohort 1b: LBL-007 + Tislelizumab + Bevacizumab + 5-Fluorouracil (5-FU) (Experimental): LBL-007 (medium dose) + tislelizumab (high dose once every 4 weeks) + bevacizumab (5 mg/kg once every 2 weeks) + 5-FU
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: 5-Fluorouracil
- Phase 1b: Cohort 2: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine (Experimental): LBL-007 (high dose) + tislelizumab (low dose every 3 weeks or high dose every 4 weeks) + bevacizumab (7.5 mg/kg once every 3 weeks or 5 mg/kg once every 2 weeks) + fluoropyrimidine (5-FU or capecitabine)
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: Capecitabine; Drug: 5-Fluorouracil
- Phase 2: Arm A and Arm D: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine (Experimental): LBL-007 (high dose) + tislelizumab (low dose every 3 weeks or high dose every 4 weeks) + bevacizumab (7.5 mg/kg once every 3 weeks or 5 mg/kg once every 2 weeks) + fluoropyrimidine (5-FU or capecitabine)
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: Capecitabine; Drug: 5-Fluorouracil
- Phase 2: Arm B: LBL-007 + Bevacizumab + Fluoropyrimidine (Experimental): LBL-007 (high dose) + bevacizumab (7.5 mg/kg once every 3 weeks or 5 mg/kg once every 2 weeks) + fluoropyrimidine (5-FU or capecitabine)
  Interventions: Drug: LBL-007; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: Capecitabine; Drug: 5-Fluorouracil
- Phase 2: Arm C and Arm E: Bevacizumab + Fluoropyrimidine (Active Comparator): Bevacizumab (7.5 mg/kg once every 3 weeks or 5 mg/kg once every 2 weeks) + fluoropyrimidine (5-FU or capecitabine)
  Interventions: Drug: LBL-007; Drug: Tislelizumab; Drug: Bevacizumab or Bevacizumab biosimilar; Drug: Capecitabine; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: LBL-007 — Administered intravenously.
  Other Names: Alcestobart
Drug: Tislelizumab — Administered intravenously.
  Other Names: BGB-A317
  Arms: Phase 1b: Cohort -1: LBL-007 + Tislelizumab + Bevacizumab + Capecitabine; Phase 1b: Cohort 1a: LBL-007 + Tislelizumab + Bevacizumab + Capecitabine; Phase 1b: Cohort 1b: LBL-007 + Tislelizumab + Bevacizumab + 5-Fluorouracil (5-FU); Phase 1b: Cohort 2: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine; Phase 2: Arm A and Arm D: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine; Phase 2: Arm C and Arm E: Bevacizumab + Fluoropyrimidine
Drug: Bevacizumab or Bevacizumab biosimilar — Administered intravenously
Drug: Capecitabine — Administered in accordance with relevant local guidelines and/or prescribing information
  Arms: Phase 1b: Cohort -1: LBL-007 + Tislelizumab + Bevacizumab + Capecitabine; Phase 1b: Cohort 1a: LBL-007 + Tislelizumab + Bevacizumab + Capecitabine; Phase 1b: Cohort 2: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine; Phase 2: Arm A and Arm D: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine; Phase 2: Arm B: LBL-007 + Bevacizumab + Fluoropyrimidine; Phase 2: Arm C and Arm E: Bevacizumab + Fluoropyrimidine
Drug: 5-Fluorouracil — Administered in accordance with relevant local guidelines and/or prescribing information
  Arms: Phase 1b: Cohort 1b: LBL-007 + Tislelizumab + Bevacizumab + 5-Fluorouracil (5-FU); Phase 1b: Cohort 2: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine; Phase 2: Arm A and Arm D: LBL-007 + Tislelizumab + Bevacizumab + Fluoropyrimidine; Phase 2: Arm B: LBL-007 + Bevacizumab + Fluoropyrimidine; Phase 2: Arm C and Arm E: Bevacizumab + Fluoropyrimidine

SUMMARY:
This is a Phase 1b/2 study to investigate the efficacy and safety of LBL-007 plus tislelizumab when administered in combination with bevacizumab plus fluoropyrimidine, and LBL-007 in combination with bevacizumab plus fluoropyrimidine versus bevacizumab plus fluoropyrimidine to participants with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have measurable disease as defined per RECIST version 1.1
* Has a histologically confirmed colorectal adenocarcinoma with metastatic or unresectable disease (Stage IV as defined by American Joint Committee on Cancer [AJCC] 8th edition)
* No prior systemic therapy for colorectal cancer (CRC) in the metastatic setting except for the induction treatment of first-line therapy. Note: Local regional treatment performed during induction systemic treatment is allowed
* Participants who have completed the first-line induction treatment, with an overall response of stable disease or better. The duration of induction treatment should be completed within approximately 6 months. The first dose of study treatment needs to occur within 2 weeks (for 2-week regimen) or 3 weeks (for 3-week regimen) to 6 weeks after Day 1 of the last cycle of induction therapy

Exclusion Criteria:

* Participants whose disease has become resectable at the investigator's discretion during or after induction treatment are not eligible
* Progressive disease occurred less than 6 months from completion of any prior neoadjuvant therapy (ie, chemotherapy with or without radiotherapy) or adjuvant therapy (ie, chemotherapy with or without radiotherapy), whichever occurred later
* Participants who have been treated with anti-epidermal growth factor receptor (EGFR) antibody in the induction treatment
* Any prior therapy targeting T-cell stimulation or checkpoint pathways
* Participants with B-raf proto-oncogene, serine/threonine kinase (BRAF)V600E mutations
* Have locally or centrally confirmed microsatellite instability-high (MSI-H) by polymerase chain reaction (PCR) method or dMMR by immunohistochemistry (IHC) method

Note: Other protocol defined criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of participants with Adverse Events (AEs) and Serious AEs (SAEs) | From the first dose of study drug(s) to 30 days after last dose, initiation of new anticancer therapy, death, withdrawal of consent, or loss to follow-up, whichever occurs first (up to approximately 28 months)
  Number of participants with AEs and SAEs characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 [NCI-CTCAE v5.0]).
Phase 2: Progression Free Survival (PFS) as Assessed by The Investigator in PD-L1 Positive Arms A and C | Approximately 28 months
  PFS, as assessed by the investigator per RECIST v1.1 is defined as the time from the date of randomization to the date of first documentation of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Phase 2: Objective Response rate (ORR) as Assessed by The Investigator in PD-L1 Positive Arms A and C and PD-L1 Negative Arms D and E | Approximately 28 months
  ORR is defined as the proportion of participants with a confirmed complete response (CR) or partial response (PR) from the time of randomization.
Phase 2: Duration of response (DOR) as Assessed by The Investigator in PD-L1 Positive Arms A and C and PD-L1 Negative arms D and E | Approximately 28 months
  DOR is defined as the time from the first confirmed objective response after randomization until the first documentation of disease progression or death, whichever comes first.
Phase 2: Progression Free Survival (PFS) as Assessed by The Investigator in PD-L1 Negative Arms D and E | Approximately 28 months
  PFS, as assessed by the investigator per RECIST v1.1 is defined as the time from the date of randomization to the date of first documentation of disease progression or death, whichever occurs first.
Phase 2: Number of participants with AEs and SAEs | From the first dose of study drug(s) to 30 days after the last dose, initiation of new anticancer therapy, death, withdrawal of consent, or loss to follow-up, whichever occurs first (up to approximately 28 months)
  Number of participants with AEs and SAEs characterized by type, frequency, severity as graded by NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (76):
- United States (30):
  - Alaska Oncology and Hematology, Llc, Anchorage, Alaska
  - Banner Md Anderson Cancer Center, Gilbert, Arizona
  - Toi Clinical Research, Cerritos, California
  - Usc Norris Comprehensive Cancer Center (Nccc), Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA, Los Angeles, California
  - Hoag Memorial Presbyterian, Newport, California
  - Kaiser Permanente Northern California, Vallejo, California
  - Baptist Md Anderson Cancer Center, Jacksonville, Florida
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Cancer Care Specialists, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Perlmutter Cancer Center At Winthrop Oncology Hematology Associatesnyu Winthrop Hospital, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center At Nyu Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Ut Southwestern Medical Center, Dallas, Texas
  - Ut Health San Antonio Mays Cancer Center, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Cancer Care Northwest, Spokane Valley, Washington
  - Multicare Health System Institute For Research and Innovation, Tacoma, Washington
- Australia (13):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Orange Health Service (Central West Cancer Care Centre), Orange, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Flinders Centre For Innovation in Cancer (Fcic), Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - St John of God, Murdoch, Murdoch, Western Australia
  - One Clinical Research, Nedlands, Western Australia
- China (32):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Quanzhou First Affliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Nanyang Central Hospital, Nanyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Nantong First Peoples Hospital, Nantong, Jiangsu
  - Affiliated Hospital of Jiangnan University South Campus, Wuxi, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jining No.1 Peoples Hospital West Branch, Jining, Shandong
  - Linyi Peoples Hospital, Linyi, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai 10Th Peoples Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital Branch Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Union Medical Center (Nankai University Affiliated Hospital), Tianjin, Tianjin Municipality
  - Karamay Central Hospital of Xinjiang, Karamay, Xinjiang
  - The Xinjiang Uygur Autonomous Region Peoples Hospital, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Pan American Oncology Trials, Llc, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/